CLINICAL TRIAL: NCT03429010
Title: Efficacy of Perioperative Anesthesia Care Bundle on Prognosis in Elderly Undergoing Hip Fracture Surgery: a Single-center Randomized Controlled Trial
Brief Title: Efficacy of Perioperative Anesthesia Care Bundle on Prognosis in Elderly Undergoing Hip Fracture Surgery
Acronym: EPAPHUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2017-03-110
Record Dates: First submitted 2018-01-18; First posted 2018-02-12 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Anesthesia; Hip Fracture Surgery; Nursing
Keywords: Anesthesia; Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New "guideline" (Experimental): New "guideline" anesthesia strategy team (Group A)
  Interventions: Procedure: New "guideline" anesthesia strategy team
- Current strategy (No Intervention): Current anesthesia strategy team (Group B)

INTERVENTIONS:
Procedure: New "guideline" anesthesia strategy team — New "guideline" anesthesia strategy team
  Arms: New "guideline"

SUMMARY:
This study is going to research the hypothesis that to strengthen the comprehensive treatment of perioperative anesthesia is possible to improve the prognosis of patients with hip fracture and reduce mortality. This is a randomized controlled pilot study aimed to elderly patients with hip fracture on one side and needing surgical treatment.

DETAILED DESCRIPTION:
To evaluate the efficacy of perioperative anesthesia care bundle on prognosis in elderly undergoing hip fracture surgery; to assess the levels of compliance that current anesthesia management strategy of our hospital against the new "guidelines"; and to analyze the defects in the current anesthesia management strategy and collect data for further multi-center research, this single-center randomized controlled trial was conducted. The central stochastic system was adopted to determined the stratification factors by age, POSSUM score, whether there was tracheal intubation or laryngeal mask auxiliary ventilation. Therefore, there are two groups including the new version of "guidelines" anesthesia strategy group and existing anesthesia strategy group at a ratio of 1:1. The mortality is the primary indicator will be collected in 1,6,12 months after surgery. And VAS score, MMSE, length of hospital stay and so forth, which would be collected as the secondary indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 75 years old;
2. Patients with hip fracture purely and surgical treatment is scheduled.

Exclusion Criteria:

1. Surgical treatment has been performed after entering hospital;
2. Multiple trauma: multiple fractures; chest, abdomen, pelvis and sacral trauma; severe head injury, etc.
3. Refuse to sign informed consent;
4. Investigator thinks he/she is inappropriate to carry out this study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 6 months after surgery
  Mortality in 6 months of postoperative

SECONDARY OUTCOMES:
Visual Analogue Score(VAS) | within two days after surgery
  The intensity of postoperative pain using Visual Analogue Score(VAS), has a total score of 10 range from 0 to 10. Do higher values represent a severer pain.
Complications | post-operation to discharge, an average of 2 weeks
  The incidence of postoperative complications
Death rate | Within 30 days and 1 year after surgery
  Mortality for postoperative of 30 days and 1 year
Survival time | up to one year after surgery
  Observed length of time after surgery to death within one year
Compliance score | Duration of hospital stay, an average of 2 weeks
  The level of compliance of new "guideline"(from the ratio of (score:total score)), the ratio from 0% to 100%
Hospital stay | Up to discharge,an average of 2 weeks
  Length of time stay in hospital
Cost | Length of hospital stay,an average of 2 weeks
  Total cost in hospital and expenditure for anesthesia
MMSE | Two days after surgery
  Cognitive function with Mini-Mental State Examination (MMSE)
Satisfaction score | Two weeks before discharge
  Overall satisfaction of patients, with a range of 0 to 5 points. 0 point represents not satisfied at all and 5 points mean greatly satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

DOCUMENTS (1):
  • Study Protocol (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03429010/Prot_000.pdf